CLINICAL TRIAL: NCT01530854
Title: Plasma Free Fatty Acids in Risk Assessment of Sepsis in the Emergency Department: A Prospective Pilot Study
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Cheetah Medical Inc. (Industry)
Responsible Party: Principal Investigator, Rakesh Engineer, Principal Investigator, The Cleveland Clinic
Other Study IDs: 07-969; 07-969 (Other: Cleveland Clinic)
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Sepsis
Keywords: sepsis; free fatty acids; emergency department
MeSH Terms: conditions — Sepsis; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (10 cc. total) are to be collected in non-heparinized tubes upon initial presentation to the ED as well as 3-6hours and 24(+/-3) hours after the initial blood draw. The 3-6hour and 24-hour blood draw will be optional depending on patient location and the availability of study personnel. The plasma samples will be aliquoted and frozen at -70°C for later assays. These samples will be assayed for plasma FFA, plasma glucose, plasma insulin, and future cytokines including IL-1 and TNF.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Septic
- Healthy

SUMMARY:
Plasma free fatty acids (FFAs) are thought to play a role in the generation of organ dysfunction. The investigators hypothesize that plasma FFA levels are a marker of poor prognosis in patients with sepsis. The present study will examine the relation between plasma FFA levels and severity of illness in patients with sepsis presenting to the Emergency Department. It will also examine the relation between plasma FFA levels and the risk of developing late morbidity, multiple organ dysfunction syndrome (MODS) and/or mortality during initial hospitalization and over a 30-day follow-up period.

DETAILED DESCRIPTION:
The long term objective of this study is to investigate the mechanism by which plasma free fatty acids (FFAs) contribute to the progression of sepsis severity in infectious patients presenting to the Emergency Department. In the present study, pilot data will be generated to validate our hypothesis that elevated free fatty acids are related to outcome in sepsis.

We will examine our hypotheses with the following specific aims:

1. To determine if plasma FFA levels are related to severity of illness in patients with sepsis presenting to the Emergency Department.
2. To study the prognostic value of plasma FFA levels at predicting future morbidity and mortality in patients with sepsis presenting to the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to provide informed consent (or has surrogate present that can do so)
* Presenting to the Emergency Department (ED) for evaluation
* Clinical suspicion of infection, as indicated by the ED physician's ordering a blood culture or a current temperature of ≥38C.

Exclusion Criteria:

* Liver disease
* Hepatitis
* Alcohol consumption >2 drinks/day for longer than 6 months
* Pregnant women
* Prisoners or other institutionalized individuals
* Unable to speak the English language
* Unwilling or unlikely to be reachable by telephone for the 30-day follow-up status assessment call

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective, specimen-procurement pilot study that will enroll adult patients (aged 18 years or older) who present to the Cleveland Clinic Emergency Department with suspected infection.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Disposition: Admission to hospital or discharge home | within 48 h
Hospital length-of-stay | 30 days

SECONDARY OUTCOMES:
All cause mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Engineer, MD, Principal Investigator — The Cleveland Clinic; Caitlin W Hicks, BA, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States